CLINICAL TRIAL: NCT04569526
Title: Ultrasonography Guided Brain Lesions Resection: a Tool for a Real Time Intraoperative Neuronavigation
Brief Title: Ultrasonography Guided Brain Lesions Resection:
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sarah Ahmed Saad, resident doctor, neurosurgery department, Assiut University
Other Study IDs: intra operative ultrasound
Record Dates: First submitted 2020-09-24; First posted 2020-09-30 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Patients Who Are Diagnosed to Have Intracranial Lesions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: use of intraoperative ultrasound — Ultrasonography guided brain lesions resection intra operatively for good localization

SUMMARY:
1. Evaluate the clinical value of intraoperative ultrasonography as a real-time guidance
2. Combination of data of MRI Tractography and intra operative ultrasonography will be useful in good localization of lesions or not .
3. Maximal safe resection .

DETAILED DESCRIPTION:
Accurate pre and intraoperative localization of Brain lesions is a challenge in neurosurgery specially deep intra cerebral lesions. Stereotaxy and neuronavigator played a major role in preoperative and intraoperative evaluation of exact location of intra cerebral lesions, the main drawbacks of using steriotaxy and neuronavigator that they are time consuming, complicated and expensive.(1) Nowadays we use MRI Tractography as preoperative imaging to localize lesions and there relation to neural tracts specially in eloquent brain areas, and also intraoperative ultrasonography Which act as a real-time, unexpansive and relatively simple tool for intraoperative visualization of the lesion's location, size, extent and its relationship with the surrounding tissue, also it can reveal the lesion's blood supply, it can measure the rate and direction of arterial blood flow.(2,3,4) Intraoperative ultrasonic imaging was first applied as a real-time navigation system in neurosurgery in 1980. (5) In this research we will combine the use of preoperative MRI tractography with intra operative ultrasonography in accurate localization of brain lesions and its relation with important tracts and if this combination will be beneficial and add to the safety of excision of lesions or not.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed to have Intracranial lesions Patients with recurrent lesions

Exclusion Criteria:

* Patients who are unfit for surgery Patients who have multifocal lesions

Ages: 1 Month to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed to have brain lesion, selected based on the inclusion and exclusion criteria
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2020-09-25 (Estimated); Primary Completion 2021-07-25 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Extent of resection of the lesion | 48 hours
  Extent of resection of the lesion evaluated by comparing pre operative and post operative MRI

SECONDARY OUTCOMES:
post operative complication | one month
  post operative complication evaluated by full neurological examination

CONTACTS AND LOCATIONS:
Overall Officials: Radwan nouby mahmoud, prof, Study Director — assuit nuiversity hospital neurosurgery department; wael mohamed ali, prof, Study Director — assuit nuiversity hospital neurosurgery department; mohamed aly ragaee, prof, Study Director — assuit nuiversity hospital neurosurgery department

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: related info — https://ejnpn.springeropen.com/articles/10.1186/s41983-019-0117-4
- See also: related info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3139346/